CLINICAL TRIAL: NCT06886139
Title: A Multicenter, Open-Label, Single-Arm, Phase 2 Study to Evaluate the Efficacy and Safety of TRS005 in Patients With CD20-Positive Relapsed or Refractory Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: A Phase 2 Study of TRS005 in Patients With CD20-positive R/R DLBCL.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Teruisi Pharmaceutical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRS00502001
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-04

CONDITIONS: CD20-positive Diffuse Large B-Cell Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TRS005 (Experimental): Recombinant anti-CD20 monoclonal antibody-MMAE conjugte for injection (TRS005). TRS005 at a dose of 1.8 mg/kg intravenously on day 1 of each 21-day cycle.
  Interventions: Drug: TRS005

INTERVENTIONS:
Drug: TRS005 — Recombinant anti-CD20 monoclonal antibody-MMAE conjugte for injection. To be used under medical supervision.

SUMMARY:
This trial is a multicenter, open-label, single-arm, Phase II Study. Patients with CD20 positive recurrent or refractory diffuse large B-cell lymphoma and had failed ≥2 prior lines of standard treatment will be recruited. The purpose of this trial is to evaluate the efficacy, safety, pharmacokinetic (PK) and immunogenicity characteristics of TRS005 via intravenous drip.

DETAILED DESCRIPTION:
The participants were screened and examined according to the protocol before enrollment. Participants received TRS005 at a dose of 1.8 mg/kg intravenously on day 1 of each 21-day cycle. The primary endpoints were objective response rate (ORR) assessed by Independent Review Committee (IRC). Participants were assessed for efficacy at the end of cycle 2, cycle 4, cycle 6 and every 4 subsequent cycles (each cycle is 21 days). Tumor responses were assessed by computerized tomography (CT) or positron emission tomography-computerized tomography (PET-CT) scanning per the Lugano 2014 criteria. The safety were assessed per the National Cancer Institute-Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years, gender is not limited.
2. The participants need to undergo pathological biopsy of tumor tissue.. Confirmed by histopathology with CD20-positive DLBCL, except for High-grade B-cell lymphoma with MYC and BCL2 rearrangements (HGBL-DH), and histologic transformed DLBCL according to the WHO 2022 revised classification standards.
3. Relapse or refractory after at least 2 lines of sufficient standard treatment regimens.
4. Not considered to be eligible for Autologous Stem Cell Transplant (ASCT).
5. Have measurable disease, including at least 1 nodal site measuring >1.5 cm or 1 extranodal site measuring >1.0 cm in longest dimension on computed tomography (CT).
6. Previously received anti-tumor treatment such as radiotherapy, biotherapy, immunotherapy at least 28 days before the first administration of this study; chemotherapy at least 21 days before the first administration of this study; hormone therapy at least 14 days before the first administration of this study.
7. Fully recovered from the acute toxic effects (except alopecia) to ≤ grade 1 (CTCAE 5.0) to prior anti-cancer therapy.
8. Organ Function Requirements：Adequate hematologic, renal, and hepatic function.
9. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
10. Participants must have a life expectancy of ≥3 months.
11. For women of childbearing potential and men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception. For women of childbearing potential, a negative serum pregnancy test result within 7 days before the first administration.
12. All participants and/or their parents or legal guardians must sign a written informed consent form.

Main Exclusion Criteria:

1. A history of drug allergy to components of the test drug, xenoproteins, biological agents, etc., or severe infusion reaction after previous monoclonal antibody treatment.
2. Serologic evidence of chronic hepatitis B virus (HBV) infection and unable or unwilling to receive standard prophylactic antiviral therapy or with detectable HBV viral load; Serologic evidence of hepatitis C virus (HCV) infection without completion of curative treatment or with detectable HCV viral load; Human immunodeficiency virus (HIV) seropositive.
3. Tumor-infiltrating diseases of the central nervous system.
4. Prior systemic treatment of lymphoma with MMAE-containing ADC drugs.
5. Prior treated with radiotherapy covering more than 30% of the bone marrow area.
6. ≥Grade 2 or greater baseline peripheral neuropathy.
7. Investigator-assessed diabetes uncontrolled by drug therapy.
8. Participants with other malignancies within the past 5 years.
9. Clinically significant third space fluid accumulation (i.e., ascites requiring drainage or pleural effusion that is either requiring drainage or associated with shortness of breath, etc.).
10. Active of autoimmune disease or immune deficiency.
11. Accompanied significant cardiovascular disease.
12. Participants who received autologous stem cell transplantation and CAR-T within 3 months prior to first administration; Participants who have received allogeneic stem cell transplantation in the past.
13. Participants must not have an uncontrolled infection.
14. Various vaccines were inoculated within 28 days prior to first administration.
15. Participate in clinical trials of other drugs or medical devices within 28 days prior to first administration.
16. Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
17. Pregnancy and/or active Breast Feeding.
18. Investigators assessed as unsuitable to participate in this study for other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
ORR, Objective Response Rate | At the end of cycle 2, cycle 4, cycle 6 and every 4 subsequent cycles (each cycle is 21 days)
  Objective Response Rate (ORR): the presence of at least one confirmed CR/PR. Independent Review Committee (IRC) confirmed ORR per Lugano 2014 criteria will be determined in the intention-to-treat (ITT) population.

SECONDARY OUTCOMES:
ORR, Objective Response Rate | At the end of cycle 2, cycle 4, cycle 6 and every 4 subsequent cycles (each cycle is 21 days)
  Investigator-assessed confirmed ORR per Lugano 2014 criteria will be determined in the intention-to-treat (ITT) population.
DCR, Disease Control Rate | At the end of cycle 2, cycle 4, cycle 6 and every 4 subsequent cycles (each cycle is 21 days)
  DCR is defined as the percentage of participants who have achieved complete response, partial response and stable disease to a therapeutic intervention. Investigator-assessed and IRC confirmed DCR per Lugano 2014 criteria.
PFS, Progression-free survival | At the end of cycle 2, cycle 4, cycle 6 and every 4 subsequent cycles (each cycle is 21 days)
  PFS is defined as the time from the start of treatment to progressive disease (PD) or death due to any cause in the absence of documented PD. Investigator-assessed and IRC confirmed PFS per Lugano 2014 criteria.
DOR, Duration of response | At the end of cycle 2, cycle 4, cycle 6 and every 4 subsequent cycles (each cycle is 21 days)
  DOR is defined as the time from the date of the first documentation of response in participants with confirmed objective tumor response (complete response or partial response) to the first documentation of progressive disease (PD) or to death due to any cause in the absence of documented PD. Investigator-assessed and IRC confirmed DOR per Lugano 2014 criteria.
TTP, Time to progression | At the end of cycle 2, cycle 4, cycle 6 and every 4 subsequent cycles (each cycle is 21 days)
  TTP is defined as the time from the start of treatment to progressive disease (PD). Investigator-assessed and IRC confirmed TTP per Lugano 2014 criteria.
OS, Overall survival | 24 months after the end of treatment in the last participant
  OS is defined as the time from the start of treatment to death due to any cause and will be analyzed by Kaplan-Meier method.
Number of Participants with Treatment-Related Adverse Events (AEs) | Through study completion, an average of 1 year
  AEs will be assigned to preferred term using MedDRA and graded according to CTCAE v5.0.
Number of Participants with Immunogenicity | At the end of cycle 2, cycle 4, cycle 6 and every 4 subsequent cycles (each cycle is 21 days)
  ADA will be assessed in all participants. NAb will be assessed in samples that are ADA positive.

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Chinese Academy of Medical Sciences, Cancer Hospital, Beijing, Beijing Municipality, China